CLINICAL TRIAL: NCT02553824
Title: Qsymia (Phentermine-topiramate) to Reduce Binge Eating/Purging in Patients With Bulimia Nervosa and Binge Eating Disorder
Brief Title: FDA Approved Medication to Reduce Binge Eating and/or Purging
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Debra L. Safer, Associate Professor, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 31390
Record Dates: First submitted 2015-08-21; First posted 2015-09-18 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Binge Eating Disorder; Bulimia Nervosa
Keywords: binge eating; bulimia nervosa; binge eating disorder; eating disorder treatment
MeSH Terms: conditions — Binge-Eating Disorder; Bulimia Nervosa; Bulimia | interventions — Phentermine; Qsymia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phentermine/Topiramate-First + Placebo (Experimental): Patients randomly assigned to this condition will receive the study medication first, have a 2 week washout, and then crossover to receive the control medication/placebo
  Interventions: Drug: Phentermine/Topiramate-First; Drug: Placebo
- Placebo-First + Phentermine/Topiramate (Placebo Comparator): Patients randomly assigned to this condition will receive the control medication (placebo) first followed by a 2 week washout, and then receive the study medication.
  Interventions: Drug: Phentermine/Topiramate-First; Drug: Placebo

INTERVENTIONS:
Drug: Phentermine/Topiramate-First — Patients randomly assigned to this Arm will have a 4 week ramp up period (in which doses will be increased, as tolerated, starting from 3.75 mg/23 mg, 7.5 mg/46 mg ,11.25 mg/69 mg , 15 mg/92 mg taken once daily in the morning. For the final 8 weeks, participants will take the 15mg/92 mg (or highest dose tolerated). Then will have a 2 week washout followed by a crossover to 12 weeks of control medication/ placebo.
  Other Names: Qsymia
Drug: Placebo — Patients randomly assigned to this Arm will have begin with 12 weeks of placebo followed by a 2 week washout. They will then crossover to Qsymia and receive a 4 week ramp up period (in which doses will be increased, as tolerated, starting from 3.75 mg/23 mg, 7.5 mg/46 mg ,11.25 mg/69 mg , 15 mg/92 mg taken once daily in the morning. For the final 8 weeks, participants will take the 15mg/92 mg (or highest dose tolerated).
  Other Names: Placebo-First

SUMMARY:
This study will demonstrate the efficacy of Qsymia versus placebo in treating bulimia nervosa and binge eating disorder.

DETAILED DESCRIPTION:
Bulimia nervosa (BN) and binge eating disorder (BED) are serious mental disorders associated with adverse psychological and physical consequences. Treatment options to date offer limited success, leaving at least 50-70% of patients still symptomatic after treatment. The purpose of the study is to evaluate whether phentermine-topiramate (Qsymia), a medication currently FDA approved for the treatment of obesity, will demonstrate efficacy-compared to placebo- when re-purposed for patients with bulimia and binge eating.

Participants will be randomized into one of two conditions: qsymia or Placebo. One condition will receive 3 months of phentermine-topiramate, a 2 week washout, then 3 months of placebo. The other condition will receive 3 months of Placebo, a 2 week washout, then 3 months of phentermine-topiramate. Participants will receive a total of 6 months of treatment and then have a 2 month follow-up off of medications.

ELIGIBILITY:
Inclusion Criteria:

* Must meet Diagnostic and Statistical Manual -Edition 5 criteria for bulimia or binge eating disorder, which has not responded to prior treatment
* Men and women between the ages of 18-60
* Must be at least normal weight (i.e. body mass index at least 21.0 or greater)
* If female of child-bearing potential, the participant must have an initial negative pregnancy test and be taking adequate birth control
* must be medically stable with no new diagnoses (medical, surgical, or psychiatric) within the past 6 months
* Must live close enough or be within commute distance of study site (Stanford, CA) to be able to comply with study visits, treatment plans, and blood draws and other possible assessments (i.e. EKG)

Exclusion Criteria:

* Any patient with bipolar disease or schizophrenia or any patient taking a mood stabilizer or antipsychotic medication within the past 3 months
* Any patient with current or past history of anorexia nervosa (i.e., with a Body mass index of < 17.5).
* Any patient with prior (within 30 days) use of Over The Counter (OTC) weight-reducing agents, herbal preparations
* Any patient who has been prescribed a medication for weight loss within the past 3 months
* Any psychological weight-loss interventions (i.e., Weight Watchers, Jenny Craig) in which patient has lost weight over the past month (unless willing to discontinue).
* Any patient currently in therapy with a psychostimulant or who has used a psychostimulant within the past 6 months
* Any patient with known sensitivity to phentermine or topiramate
* Any patient who has had a change in thyroid, psychiatric, or blood pressure medications within the past one month
* Any patient who is taking a potassium-wasting diuretic
* Any patient who is on a carbonic anhydrase inhibitor such as zonisamide acetazolamide, or dichlorphenamide
* Any diabetic who is taking insulin or an insulin secretagogue
* Any patient with liver enzymes at baseline greater than three times the upper limit of normal
* Any patient with a baseline potassium of less than 3.0 millequivalent/Liter. Patients with baseline potassium levels between 3.0-3.5 miliEquivalents/Liter will be encouraged to ingest high potassium foods such as bananas, oranges, or tomato juice daily during the study
* Any patient with abnormal baseline thyroid test or with a Thyroid Stimulating Hormone (TSH) greater than 1.5 times the upper limit of normal
* Any patient who is unwilling or expresses uncertainty about being able to refrain from daily alcohol use (even if at moderate levels) or illegal drugs while taking the study medication.
* Any adult with recent history of suspected alcohol or substance abuse or substance dependence
* Any patient who regularly uses marijuana (including medical marijuana) or illegal drugs
* Any patient who has a history of addiction to a stimulant
* Any patient who expresses current suicidal ideation
* Any patient with a history of nephrolithiasis
* Any patient who is pregnant or who is planning to become pregnant during the study period.
* Any patient who is currently participating in any other clinical study that involves an active treatment
* Any patient who is unable to identify a primary care physician
* Any patient with a history of cardiovascular disease (i.e. recent history of Myocardial Infarction, stroke, shortness of breath, chest pain) that could increase vulnerability to the sympathomimetic effects of a stimulant like drug. If clinical suspicion is high, baseline EKG will be obtained and anyone with abnormal findings will be excluded

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2015-10-30 (Actual); Primary Completion 2017-02-23 (Actual); Study Completion 2017-04-15 (Actual)

PRIMARY OUTCOMES:
Frequency of binge eating episodes as measured by the Eating Disorder Examination Assessment | 8.5 months
  The primary outcome is the frequency of binge episodes

SECONDARY OUTCOMES:
Frequency of binge eating episodes measured by the Eating Disorder Examination Assessment | 8.5 months
  Frequency of binge episodes
Percentage of Abstinence from Binge Eating as Measured by the Eating Disorder Examination Assessment | 8.5 months
  Percentage of patients who have had no binge episodes as assessed by the EDE

CONTACTS AND LOCATIONS:
Overall Officials: Debra L Safer, MD, Principal Investigator — Stanford University; Sarah Adler, PsyD, Principal Investigator — Stanford University; Shebani Sethi, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford School of Medicine, Psychiatry and Behavioral Sciences, Stanford, California, United States

REFERENCES:
- [Derived] Safer DL, Adler S, Dalai SS, Bentley JP, Toyama H, Pajarito S, Najarian T. A randomized, placebo-controlled crossover trial of phentermine-topiramate ER in patients with binge-eating disorder and bulimia nervosa. Int J Eat Disord. 2020 Feb;53(2):266-277. doi: 10.1002/eat.23192. Epub 2019 Nov 13. PMID 31721257
- [Derived] Dalai SS, Adler S, Najarian T, Safer DL. Study protocol and rationale for a randomized double-blinded crossover trial of phentermine-topiramate ER versus placebo to treat binge eating disorder and bulimia nervosa. Contemp Clin Trials. 2018 Jan;64:173-178. doi: 10.1016/j.cct.2017.10.007. Epub 2017 Oct 14. PMID 29038069